CLINICAL TRIAL: NCT07209267
Title: Baricitinib Curative Repression of HIV-1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Vincent Marconi, Professor of Medicine, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00009759; 2025P012728 (Other: Emory IRB)
Record Dates: First submitted 2025-10-02; First posted 2025-10-06 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: HIV Infection; HIV
Keywords: Baricitinib; Antiretroviral Therapy (ART)
MeSH Terms: conditions — HIV Infections | interventions — Antiretroviral Therapy, Highly Active; Standard of Care; baricitinib

STUDY DESIGN:
Intervention Model Description: Step 1: Participants with well-controlled HIV on ART will be treated for 26 weeks with baricitinib 2 plus their current ART regimen.
  Step 2: Following 26 weeks of baricitinib plus ART, participants will be treated with baricitinib alone (ART will be interrupted) for up to 24 weeks.
  Step 3: Participants should return as soon as possible after an ART restart criterion has been met or at the end of Step 2. Participants will be followed for 24 weeks during this step.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Baricitinib (Experimental): Adults with well-controlled HIV on ART will be treated for 26 weeks with baricitinib 2 mg per day orally plus their current ART regimen (Step 1).
  Following 26 weeks of baricitinib plus ART, ART will be interrupted, and the participants will be treated with baricitinib alone for up to 24 weeks (Step 2).
  If a participant qualifies for ART restart criteria before the end of the maximum 24 weeks of Step 2, they will move to Step 3 early and resume ART, while baricitinib will be discontinued for 24 weeks. Otherwise, participants will remain on baricitinib alone until the end of the 24 weeks of Step 2 and will then resume ART while baricitinib is discontinued for an additional 24 weeks of observation (Step 3).
  Interventions: Drug: Antiretroviral Therapy (ART); Drug: Baricitinib (LY3009104) 2 mg

INTERVENTIONS:
Drug: Antiretroviral Therapy (ART) — Antiretroviral Therapy (ART): A treatment regimen for HIV infection that uses a combination of antiretroviral drugs to suppress viral replication, reduce HIV-related morbidity, and prevent transmission.
  In Step 1, participants will continue their current ART regimen for 26 weeks.
  In Step 2, participants will interrupt ART.
  In Step 3, participants will restart ART treatment early if they meet the ART restart criteria before the end of Step 2 (24-week maximum). Otherwise, they will resume ART at the end of Step 2.
  Other Names: Standard of Care
Drug: Baricitinib (LY3009104) 2 mg — Baricitinib is an orally administered, selective inhibitor of Janus kinase (JAK) 1 and 2. It reduces cytokine-mediated signaling involved in inflammation and immune activation. Baricitinib is FDA-approved for rheumatoid arthritis (RA), atopic dermatitis, and alopecia areata. It has also been authorized for the treatment of COVID-19 in hospitalized patients.
  During Step 1, Baricitinib will be taken at a dose of 2 mg orally daily for 26 weeks.
  During Step 2, Baricitinib alone will be continued at a dose of 2 mg orally daily for up to an additional 24 weeks
  Other Names: Olumiant

SUMMARY:
This study is being done to test whether a drug called baricitinib, which blocks specific causes of inflammation, affects HIV-1 viral rebound and viral load levels after HIV treatment is discontinued. Researchers will test the effects of continuing baricitinib in people with HIV before and after discontinuing their antiretroviral therapy. This drug is approved by the Food and Drug Administration (FDA) for other diseases; it is not approved for the treatment of HIV-1. The study team will also investigate any side effects associated with the drug.

DETAILED DESCRIPTION:
This study will test whether the medication baricitinib, which reduces inflammation and is already approved for other diseases, can delay the return of HIV after stopping antiretroviral therapy (ART). The goal is to see if baricitinib can safely reduce inflammation and the HIV that is hidden in the body. The study will include adults with HIV who have a suppressed viral load on ART.

Participants will receive ART combined with baricitinib for 26 weeks, followed by baricitinib alone after stopping ART. If the virus returns, the previous ART will be restarted. Each participant will be involved in the study for approximately 12 to 18 months.

Blood and other biological samples may be stored for future research use, with the participant's consent.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* On continuous ART for at least 96 weeks before enrollment, with no interruption of ART for 7 consecutive days or longer in the 48 weeks before enrollment.
* Plasma HIV-1 RNA levels of <50 copies/mL for at least 96 weeks (a minimum of two measures), and <50 copies/mL for a sample obtained within 90 days, before enrollment.
* CD4+ T-cell count ≥500 cells/mm3 obtained within 90 days prior to enrollment
* No known history of CD4+ T-cell count nadir <200 cells/mm3
* Negative pregnancy test at time of study enrollment
* Additional laboratory criteria may apply.

Exclusion Criteria:

* < 18 years of age or > 70 years of age
* Pregnancy or breastfeeding, as determined by a blood pregnancy test
* History of AIDS-defining illness, except for recurrent pneumonia.
* History of progressive multifocal leukoencephalopathy or clinically significant HIV-associated neurocognitive disease.
* Untreated latent tuberculosis infection (which will be screened for before entry). If there is a prior positive test, the test does not need to be repeated at screening.
* History of use of any immunomodulatory medications within 6 months before enrollment, including systemic corticosteroids (>14 days), immunosuppressants, anti-cancer, interleukins, systemic interferons, systemic chemotherapy, or other medications that the site investigator feels could have an immunomodulatory effect.
* History of deep venous thrombosis
* Cardiovascular disease (Coronary artery disease or history of myocardial infarction, Congestive heart failure with left ventricular ejection fraction ≤40% per American Heart Association guidelines, history of stroke)
* History of HIV-associated malignancy, including Kaposi's sarcoma, or any lymphoma/leukemia or virus-associated cancers. Active or recent non-HIV-associated malignancy requiring systemic chemotherapy or surgery in the preceding 36 months
* Major surgery within 8 weeks before screening, or will require major surgery during the study
* Current or recent (<4 weeks before screening) clinically serious viral (including COVID-19), bacterial, fungal, or parasitic infection or any other active or recent infection. History of untreated syphilis infection. If a rapid plasma reagin (RPR) test was negative in the 3 months before screening, then an RPR is not needed at screening
* Symptomatic herpes simplex at the time of screening.
* Symptomatic herpes zoster infection within 12 weeks before screening.
* History of disseminated/complicated herpes zoster (for example, ophthalmic zoster or central nervous system (CNS) involvement).
* Positive test for hepatitis B virus (HBV)
* Additional exclusion criteria apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Time to restart ART | Up to 24 weeks after the baricitinib treatment alone was started
  Time to restart ART will be defined by a plasma HIV-1 RNA viral load greater than or equal to 1000 copies/mL following withdrawal of ART during 24 weeks of baricitinib treatment alone (following 26 weeks of baricitinib plus ART).
Number of Participants who discontinued treatment due to adverse events | Up to 24 weeks after the start of baricitinib alone was started
  Participants who permanently discontinued study drug due to treatment-related adverse events.
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | Up to 24 weeks after the start of baricitinib alone was started
  Number of participants experiencing treatment-emergent adverse events (TEAEs), including serious adverse events.

SECONDARY OUTCOMES:
Time to a detectable plasma HIV-1 RNA viral load | Up to 24 weeks after baricitinib alone was started.
  Time to a detectable plasma HIV-1 RNA viral load (defined as greater than the lower limit of quantification) after analytic treatment Interruption (ATI).

OTHER OUTCOMES:
Latent intact HIV reservoir | Baseline and up to 24 week after baricitinib alone was started.
  Latent intact HIV reservoir as measured in peripheral blood primarily by Intact Proviral DNA Assay (IPDA), integrated HIV-1 DNA (Alu-PCR), cell-associated RNA, and proviral DNA (total HIV cell-associated DNA).

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Marconi, MD, Principal Investigator — Emory University; William Tyor, MD, Principal Investigator — Emory University; Christina Gavegnano, PhD, Principal Investigator — Emory University; Andrew H Miller, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Infectious Diseases Clinic (Ponce Center), Atlanta, Georgia
  - Dr. Gavegnano's Laboratory, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
The research team will share the data that underline the results reported in articles, after deidentification
Supporting Information: Study Protocol
Time Frame: Data will be shared by the research team after the study has been completed.
Access Criteria: Requests should be sent directly to the PI via email, summarizing the purpose of utilizing the data.